CLINICAL TRIAL: NCT01492829
Title: Development and Evaluation of a Community Health Worker Delivered HIV/STI Prevention Intervention for Women Living in Internally Displaced Persons Camps in Leogane, Haiti
Brief Title: A Community-health Worker Delivered HIV/STI Prevention Intervention for Internally Displaced Women in Leogane, Haiti
Acronym: FASY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: NEGES Foundation, Leogane, Haiti (Unknown); Adelphi University (Other)
Responsible Party: Principal Investigator, Carmen Logie, Post-doctoral Fellow, Women's College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GCC#0016-01-04-01-01
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Risk Reduction Behavior; Interpersonal Relations; Mental Disorders
Keywords: HIV prevention; sexually transmitted infection prevention; HIV knowledge; relationship power; depression; coping; social support; internally displaced persons; community health worker; HIV/STI educational video; substance use; women's health
MeSH Terms: conditions — Risk Reduction Behavior; Mental Disorders; Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: individual and group-based, community health worker delivered — Pre-test will be individual, tablet-based; participants will receive correct information for incorrect HIV/STI knowledge responses and will watch a brief HIV/STI educational video. This will be followed by participants attending 6 weeks of group educational sessions focused on: HIV, STI, interpersonal relationships, communication and decision-making, mental health and coping, creating social change

SUMMARY:
The investigators will develop, deliver and evaluate a solar powered tablet-based individual and group focused HIV/STI prevention intervention with internally displaced women in Leogane, Haiti. Internally displaced women will be trained as community health workers to deliver the HIV/STI prevention intervention to other internally displaced women.

DETAILED DESCRIPTION:
We will develop and field test a multi-component intervention that includes (1) solar-powered tablets with brief video-based educational messages and (2) 6 weekly peer-group sessions. The tablet will be programmed to analyze the data and to indicate incorrect HIV knowledge responses so the community health worker can immediately provide correct responses. This intervention involves 6 weekly women's health meetings that will cover a variety of issues pertinent to women's sexual health: HIV/AIDS, sexually transmitted infections, interpersonal relationships, communication and decision making, mental health and coping, creating social change.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over
* capable of providing informed consent
* internally displaced (living in tent or camp)
* female

Exclusion Criteria:

* male
* under 18 years old
* not able to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
HIV Knowledge | 8 weeks
  Brief HIV Knowledge Questionnaire (Carey & Schroder, 2002)

SECONDARY OUTCOMES:
Sexually Transmitted Infection Knowledge | 8 weeks
  Measured using Sexually Transmitted Disease Knowledge Questionnaire (Jaworski & Carey, 2007)
Condom use | 8 weeks
  Measured using a self-report of frequency of condom use with regular, casual and paid sex sexual partners
Substance use | 8 weeks
  Measured using self-reported frequency of drug/alcohol use
Depression | 8 weeks
  Measured using Patient Health Questionnaire 2 (PHQ-2)
Social support | 8 weeks
  Measured using Multi-dimensional scale of perceived social support (Zimet et al., 1988)
resilient coping | 8 weeks
  Measured using Brief Resilient Coping Scale (Sinclair & Wallston, 2004)
Relationship Control | 8 weeks
  Sexual Relationship Power Scale (Pulerwitz, Gortmaker & DeJong, 2000)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen H Logie, PhD, Principal Investigator — Women's College Hospital
Locations (1):
- NEGES, Léogâne, Haiti

REFERENCES:
- [Derived] Logie CH, Daniel C, Wang Y. Factors associated with consistent condom use among internally displaced women in Leogane, Haiti: results from a cross-sectional tablet-based survey. Sex Transm Infect. 2016 Nov;92(7):520-524. doi: 10.1136/sextrans-2015-052400. Epub 2016 Mar 31. PMID 27034426
- [Derived] Logie CH, Daniel C, Newman PA, Weaver J, Loutfy MR. A psycho-educational HIV/STI prevention intervention for internally displaced women in Leogane, Haiti: results from a non-randomized cohort pilot study. PLoS One. 2014 Feb 28;9(2):e89836. doi: 10.1371/journal.pone.0089836. eCollection 2014. PMID 24587068
- [Derived] Logie CH, Daniel C, Newman PA, Loutfy MR. An HIV/STI prevention intervention for internally displaced women in Leogane, Haiti: study protocol for an N-of-1 pilot study. BMJ Open. 2012 Jul 18;2(4):e001634. doi: 10.1136/bmjopen-2012-001634. Print 2012. PMID 22815471